CLINICAL TRIAL: NCT06889480
Title: MultitArget STereotactic Electrophysiological Recording and Stimulation for Tourette Syndrome
Acronym: MASTERS-TS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Jianguo Zhang, Director of Department of Functional Neurosurgery, Beijing Tiantan Hospital, Capital Medical University, Beijing, China, Beijing Tiantan Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HX-B-2024057
Record Dates: First submitted 2025-03-16; First posted 2025-03-21 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-03

CONDITIONS: Tourette Syndrome; Deep Brain Stimulation
Keywords: Tourette syndrome; Electrophysiology; Tics; Psychiatric Comorbidities; Deep Brain Stimulation; Biomarker
MeSH Terms: conditions — Tourette Syndrome; Tics

STUDY DESIGN:
Intervention Model Description: This study employs a randomized crossover design. In the initial phase, each participant is randomly assigned to receive one of three different stimulation interventions - new target stimulation, CM-DBS, and sham stimulation - each for one month in a randomized order. Following this phase, the best target stimulation and short-term efficacy parameters are individually re-optimized for an additional three months to evaluate long-term efficacy. This design allows each participant to serve as their own control, thereby reducing inter-subject variability and improving the precision of treatment comparisons. Outcome measures, including tic severity and standard neuropsychiatric assessments, are administered at baseline, 1 month after each randomized stimulation period during the crossover phase, and 3 months after continuous optimal stimulation.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are blinded to the stimulation condition (i.e., whether they receive new target stimulation, CM-DBS, or sham stimulation), and the outcomes assessors are also blinded to the intervention assignments. However, due to the nature of the procedure, care providers and investigators are not masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- New Target DBS (Experimental): Participants in this arm will receive active deep brain stimulation targeted to a novel brain region. The new target is identified through electrophysiological brain mapping and 24-hour stimulation. Stimulation parameters (frequency, voltage, pulse width) will be individually optimized based on mapping results.
  Interventions: Device: New Target DBS
- CM-DBS (Active Comparator): Participants in this arm will receive active deep brain stimulation at the central medial thalamic nucleus (CM), a well-established target for TS treatment. Stimulation settings are determined during electrophysiological brain mapping and 24-hour stimulation. This arm serves as the active comparator, enabling the evaluation of relative efficacy and safety between the conventional CM target and the new target intervention.
  Interventions: Device: CM-DBS
- Sham Stimulation (Sham Comparator): Participants in this arm will undergo identical surgical procedures and follow-up assessments as in the active stimulation arms but will receive sham (inactive) stimulation. This arm is designed to control for placebo effects and ensure that any observed improvements in TS symptoms are attributable to the active interventions.
  Interventions: Device: Sham Stimulation

INTERVENTIONS:
Device: New Target DBS — Participants in this arm will receive active DBS targeting a novel brain region identified via electrophysiological brain mapping. A DBS electrode will be implanted at the new target, and stimulation parameters (including frequency, voltage, and pulse width) are individually optimized based on mapping and 24-hour testing. The procedure is performed using a robotic system for precise electrode placement, and the device is provided by Beijing PINS Medical Co., Ltd.
  Arms: New Target DBS
Device: CM-DBS — This intervention involves active DBS at the central medial thalamic nucleus (CM) -a widely used target in TS treatment. A DBS electrode is implanted at the CM target, with stimulation settings determined through electrophysiological brain mapping and subsequent 24-hour stimulation. This arm serves as an active comparator, with stimulation administered during a 1-month period in the crossover phase. The same device and robotic-assisted implantation are used to ensure consistency and precision.
  Arms: CM-DBS
Device: Sham Stimulation — Participants assigned to the sham stimulation arm undergo the identical surgical procedure and electrode implantation as those in the active arms. However, during the stimulation periods, the device is programmed to deliver no active stimulation. This sham intervention is designed to control for placebo effects and ensure that any observed improvements in TS symptoms are attributable to the active DBS interventions.
  Arms: Sham Stimulation

SUMMARY:
The goal of this clinical trial is to investigate the neural mechanisms underlying Tourette syndrome (TS) and see if personalized deep brain stimulation (DBS) can help reduce tics in TS patients and improve related issues like anxiety, attention problems, and obsessive-compulsive behaviors.

In this study, researchers will use stereoelectroencephalography (SEEG) and electrocorticography (ECoG) to record brain activity in key areas involved in movement and emotion, including the nucleus accumbens (NAc), anterior limb of the internal capsule (ALIC), insular cortex, anterior cingulate cortex (ACC), central medial thalamic nucleus (CM), globus pallidus internus (GPi), and motor cortex (M1). They will test stimulation in these areas to evaluate acute therapeutic effect for each target and to identify a new effective new target.

Later, participants will receive DBS treatment under three different conditions, each for 1 month to identify the optimal target:

1. Stimulation at the new target,
2. Stimulation at the CM,
3. Sham stimulation (does not actually stimulate).

Finally, DBS will be continued at the optimal target for an additional three months to confirm its therapeutic impact.

By analyzing the brain activity and comparing these conditions, the study will clarify the neural mechanisms underlying TS and learn which target works best to lower tics and improve overall quality of life for TS patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 60 years.
2. Diagnosis of Tourette Syndrome according to DSM-V criteria, defined as:

   i. The presence of multiple motor tics and at least one vocal tic at some point (not necessarily simultaneous).

   ii. Tics that have persisted for more than 1 year from their onset.

   iii. Onset of tics occurring before the age of 18.

   iv. The disorder is not attributable to the physiological effects of a substance or another medical condition.
3. A Yale Global Tic Severity Scale (YGTSS) total score greater than 35 (on a scale of 0-50) for at least 1 year, with a motor tic score of ≥15, and tics being the primary cause of disability.
4. Inadequate response to conservative treatments (standard pharmacological and behavioral therapy).
5. Disease duration of more than 1 year.
6. Any coexisting medical, neurological, or psychiatric disorders have been treated and remain stable for at least 6 months.
7. A stable psychosocial environment.
8. Neuropsychological evaluation demonstrating that the candidate can tolerate the surgical procedure, postoperative follow-up, and potential adverse events.
9. The participant, or his/her legal representative, is able to provide written informed consent.

Exclusion Criteria:

1. Presence of suicidal risk, defined as a score of ≥3 on the suicide-related items of the Hamilton Depression Rating Scale (HAMD).
2. History of drug or alcohol dependence within the past 6 months.
3. Abnormal brain structure as indicated by CT or MRI scans.
4. Presence of any condition that could lead to surgical failure or interfere with postoperative management.
5. Diagnosis of factitious disorder, malingering, or psychogenic tics.
6. Contraindications to neurosurgical procedures (e.g., history of cerebral infarction, hydrocephalus, cerebral atrophy, or post-stroke sequelae).
7. Contraindications for CT/MRI scanning (e.g., claustrophobia).
8. Pregnancy or lactation, or a positive pregnancy test prior to randomization.
9. Contraindications to general anesthesia (e.g., severe arrhythmia, severe anemia, hepatic or renal dysfunction).
10. Expected survival of less than 12 months.
11. Participation in other interventional clinical studies that may influence outcome assessments.
12. Any other condition that, in the investigator's judgment, renders the candidate unsuitable for participation or poses a significant risk (e.g., inability to understand study procedures or poor adherence).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in Yale Global Tic Severity Scale (YGTSS) Score | administered at baseline, 1 month after each randomized stimulation period during the crossover phase, and 3 months after continuous optimal stimulation
  The YGTSS is a 10-item semi-structured clinician-rating instrument that evaluates motor and phonic symptoms' number, frequency, intensity, complexity, and interference. The items about the tic ratings are scored on two subscales: motor tics and phonic tics. Behaviors are rated on a 6-point scale. The Total Tic Severity Score ranges from 0-50, with a higher score indicating a higher severity of symptoms.

SECONDARY OUTCOMES:
Change in Modified Rush Video Rating Scale (MRVRS) | administered at baseline, 1 month after each randomized stimulation period during the crossover phase, and 3 months after continuous optimal stimulation
  The Modified Rush Video Rating Scale (MRVRS) is a validated, video-based instrument for objectively assessing tic severity in patients with Tourette Syndrome. The MRVRS evaluates motor and phonic tics using a revised scoring method that captures tic frequency, intensity, and complexity from a 5-minute video recording. The MRVRS ranges from 0-20, with a higher score indicating a higher severity of symptoms. In this study, trained, blinded evaluators will rate each participant's tic severity using the MRVRS at multiple time points. Assessments are performed at baseline, after 1 month of stimulation during each randomized crossover period (following New Target DBS Stimulation, CM DBS Stimulation, and Sham Stimulation), and again after 3 months of continuous optimal stimulation. A decrease in the MRVRS score from baseline will indicate an improvement in tic severity.
Change in Premonitory Urge Scale (PUTS) Score | administered at baseline, 1 month after each randomized stimulation period during the crossover phase, and 3 months after continuous optimal stimulation
  The Premonitory Urge Scale (PUTS) is a self-reported measure that evaluates the intensity of premonitory urges preceding tics in patients with Tourette Syndrome. The PUTS score ranges from 9-36, where higher values reflect more severe urges, will be recorded at baseline, after each 1-month stimulation period during the randomized crossover phase, and after 3 months of continuous optimal stimulation. Changes in the PUTS score will indicate alterations in the severity of premonitory urges.
Change in Yale-Brown Obsessive Compulsive Scale (Y-BOCS) score | administered at baseline, 1 month after each randomized stimulation period during the crossover phase, and 3 months after continuous optimal stimulation
  The Yale-Brown Obsessive Compulsive Scale (Y-BOCS) is a clinician-rated instrument that assesses the severity of obsessive-compulsive disorder (OCD). Scores range from 0 (no symptoms) to 40 (severe symptoms). Assessments will be performed at baseline, after each 1-month randomized stimulation phase (following New Target DBS, CM DBS, and Sham stimulation), and after 3 months of continuous optimal stimulation. A reduction in the Y-BOCS score indicates an improvement in OCD symptoms.
Change in Conners' Adult ADHD Rating Scale (CAARS) score | administered at baseline, 1 month after each randomized stimulation period during the crossover phase, and 3 months after continuous optimal stimulation
  The Conners' Adult ADHD Rating Scale (CAARS) will be used to evaluate the severity of attention deficit hyperactivity disorder (ADHD) , including inattention, hyperactivity, and impulsivity. The scale provides a score reflecting overall ADHD severity. Assessments will be conducted at baseline, after each 1-month stimulation period during the randomized crossover phase, and after 3 months of continuous optimal stimulation. A decrease in the CAARS score indicates improvement in ADHD symptoms
Change in Hamilton Anxiety Scale (HAMA) Score | administered at baseline, 1 month after each randomized stimulation period during the crossover phase, and 3 months after continuous optimal stimulation
  The Hamilton Anxiety Scale (HAMA) is a clinician-rated scale used to assess the severity of anxiety symptoms, with scores ranging from 0 to 56. Higher scores indicate greater anxiety. HAMA assessments will be performed at baseline, after each 1-month stimulation period during the randomized crossover phase, and after 3 months of continuous optimal stimulation. A reduction in the HAMA score reflects a decrease in anxiety symptoms.
Change in Hamilton Depression Scale (HAMD) score | administered at baseline, 1 month after each randomized stimulation period during the crossover phase, and 3 months after continuous optimal stimulation
  The Hamilton Depression Scale (HAMD) is used to assess the severity of depressive symptoms, with total scores ranging from 0 to 52. Higher scores indicate more severe depression. Evaluations will occur at baseline, after each 1-month stimulation period during the randomized crossover phase, and after 3 months of continuous optimal stimulation. A reduction in the HAMD score indicates an improvement in depressive symptoms.
Change in Young Mania Rating Scale (YMRS) score | administered at baseline, 1 month after each randomized stimulation period during the crossover phase, and 3 months after continuous optimal stimulation
  The Young Mania Rating Scale (YMRS) is a clinician-administered instrument assessing the severity of manic symptoms, with scores ranging from 0 to 60. Higher scores indicate more severe mania. YMRS evaluations will be performed at baseline, after each 1-month stimulation period during the randomized crossover phase, and after 3 months of continuous optimal stimulation. A reduction in the YMRS score signifies an improvement in manic symptoms.
Change in Columbia Suicide Severity Rating Scale (C-SSRS) | administered at baseline, 1 month after each randomized stimulation period during the crossover phase, and 3 months after continuous optimal stimulation
  The Columbia Suicide Severity Rating Scale (C-SSRS) primarily evaluates the presence, severity, and frequency of suicidal ideation and behaviors rather than providing a single numerical range. Typically, higher scores indicate greater suicide risk, with severity rated individually per item rather than summed into a total score. The C-SSRS will be administered at baseline, after each 1-month stimulation period during the randomized crossover phase, and after 3 months of continuous optimal stimulation. A reduction in the C-SSRS score indicates an improvement in suicidal risk.
Change in Mini-Mental State Examination (MMSE) score | administered at baseline, 1 month after each randomized stimulation period during the crossover phase, and 3 months after continuous optimal stimulation
  The Mini-Mental State Examination (MMSE) is a clinician-administered test that evaluates overall cognitive function. The MMSE provides a score ranging from 0 to 30, with lower scores indicating greater cognitive impairment. In this study, trained evaluators will assess the MMSE score at baseline, 3 months post-intervention, and 6 months post-intervention. The primary measure is the change in the MMSE score from baseline, which will reflect any improvement or decline in cognitive function due to the interventions.
Change in Montreal Cognitive Assessment Beijing Version (MoCA) score | administered at baseline, 1 month after each randomized stimulation period during the crossover phase, and 3 months after continuous optimal stimulation
  The Montreal Cognitive Assessment Beijing Version (MoCA) is a brief screening tool that evaluates multiple cognitive domains, including memory, executive function, attention, language, and visuospatial abilities. The MoCA yields a total score from 0-30, with lower scores indicating more significant cognitive deficits. In this study, the MoCA will be administered by trained evaluators at baseline, 3 months post-intervention, and 6 months post-intervention. The outcome measure is the change in the MoCA score from baseline, which will help determine the effect of the interventions on cognitive performance.
change in Gilles de la Tourette Syndrome Quality of Life Scale (GTS-QOL) score | administered at baseline, 1 month after each randomized stimulation period during the crossover phase, and 3 months after continuous optimal stimulation
  Quality of life will be evaluated using the Gilles de la Tourette Syndrome Quality of Life Scale (GTS-QOL), a patient-reported measure that assesses the impact of TS on daily functioning and overall well-being. The scale yields a total score ranging from 0-108 where lower scores indicate a better quality of life. Assessments will be performed at baseline, after each 1-month randomized stimulation phase during the crossover period, and following 3 months of continuous optimal stimulation. A decrease in the GTS-QOL score from baseline indicates an improvement in quality of life.
Incidence of Treatment-Related Adverse Events | administered at baseline, 1 month after each randomized stimulation period during the crossover phase, and 3 months after continuous optimal stimulation
  Safety will be evaluated by recording the incidence, severity, and nature of treatment-related adverse events (AEs), including surgical complications, stimulation-related side effects, and device-related issues. Data will be collected at every follow-up visit and monitored throughout the study. This measure will provide an overall safety profile of the interventions.

OTHER OUTCOMES:
New Stimulation Target Identification | administered at baseline, 1 month after each randomized stimulation period during the crossover phase, and 3 months after continuous optimal stimulation
  This outcome measure assesses the effectiveness of electrophysiological brain mapping (using SEEG) in identifying a novel stimulation target. Success is defined as the reliable identification of a new target based on electrophysiological criteria during brain mapping and subsequent 24-hour stimulation. The proportion of patients with a successfully identified new target will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Jianguo Zhang, M.D., Ph.D., Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martinez-Ramirez D, Jimenez-Shahed J, Leckman JF, Porta M, Servello D, Meng FG, Kuhn J, Huys D, Baldermann JC, Foltynie T, Hariz MI, Joyce EM, Zrinzo L, Kefalopoulou Z, Silburn P, Coyne T, Mogilner AY, Pourfar MH, Khandhar SM, Auyeung M, Ostrem JL, Visser-Vandewalle V, Welter ML, Mallet L, Karachi C, Houeto JL, Klassen BT, Ackermans L, Kaido T, Temel Y, Gross RE, Walker HC, Lozano AM, Walter BL, Mari Z, Anderson WS, Changizi BK, Moro E, Zauber SE, Schrock LE, Zhang JG, Hu W, Rizer K, Monari EH, Foote KD, Malaty IA, Deeb W, Gunduz A, Okun MS. Efficacy and Safety of Deep Brain Stimulation in Tourette Syndrome: The International Tourette Syndrome Deep Brain Stimulation Public Database and Registry. JAMA Neurol. 2018 Mar 1;75(3):353-359. doi: 10.1001/jamaneurol.2017.4317. PMID 29340590
- [Background] Muller-Vahl KR, Szejko N, Saryyeva A, Schrader C, Krueger D, Horn A, Kuhn AA, Krauss JK. Randomized double-blind sham-controlled trial of thalamic versus GPi stimulation in patients with severe medically refractory Gilles de la Tourette syndrome. Brain Stimul. 2021 May-Jun;14(3):662-675. doi: 10.1016/j.brs.2021.04.004. Epub 2021 Apr 18. PMID 33857664
- [Background] Schuller T, Gruendler TOJ, Smith EE, Baldermann JC, Kohl S, Fischer AG, Visser-Vandewalle V, Ullsperger M, Kuhn J, Huys D. Performance monitoring in obsessive-compulsive disorder: Insights from internal capsule/nucleus accumbens deep brain stimulation. Neuroimage Clin. 2021;31:102746. doi: 10.1016/j.nicl.2021.102746. Epub 2021 Jun 29. PMID 34229156
- [Background] Xiong B, Li B, Wen R, Gao Y, Gong F, Li D, Xu Y, Deng H, Xiao L, Yin S, Zhang W, Lozano AM, Wang W. Use of differential stimulation of the nucleus accumbens and anterior limb of the internal capsule to improve outcomes of obsessive-compulsive disorder. J Neurosurg. 2023 May 26;139(5):1376-1385. doi: 10.3171/2023.4.JNS221824. Print 2023 Nov 1. PMID 37243560
- [Background] McGovern RA, Sheth SA. Role of the dorsal anterior cingulate cortex in obsessive-compulsive disorder: converging evidence from cognitive neuroscience and psychiatric neurosurgery. J Neurosurg. 2017 Jan;126(1):132-147. doi: 10.3171/2016.1.JNS15601. Epub 2016 Apr 1. PMID 27035167
- [Background] O'Neill J, Piacentini JC, Peterson BS. Cingulate role in Tourette syndrome. Handb Clin Neurol. 2019;166:165-221. doi: 10.1016/B978-0-444-64196-0.00011-X. PMID 31731911
- [Background] Jackson SR, Sigurdsson HP, Dyke K, Condon M, Jackson GM. The role of the cingulate cortex in the generation of motor tics and the experience of the premonitory urge-to-tic in Tourette syndrome. J Neuropsychol. 2021 Sep;15(3):340-362. doi: 10.1111/jnp.12242. Epub 2021 Mar 27. PMID 33774919
- [Background] Jackson SR, Loayza J, Crighton M, Sigurdsson HP, Dyke K, Jackson GM. The role of the insula in the generation of motor tics and the experience of the premonitory urge-to-tic in Tourette syndrome. Cortex. 2020 May;126:119-133. doi: 10.1016/j.cortex.2019.12.021. Epub 2020 Jan 22. PMID 32070809
- [Background] Neumann WJ, Huebl J, Brucke C, Lofredi R, Horn A, Saryyeva A, Muller-Vahl K, Krauss JK, Kuhn AA. Pallidal and thalamic neural oscillatory patterns in tourette's syndrome. Ann Neurol. 2018 Oct;84(4):505-514. doi: 10.1002/ana.25311. Epub 2018 Oct 4. PMID 30112767
- [Background] Gunduz A, Okun MS. A Review and Update on Tourette Syndrome: Where Is the Field Headed? Curr Neurol Neurosci Rep. 2016 Apr;16(4):37. doi: 10.1007/s11910-016-0633-x. PMID 26936259
- [Background] Cagle JN, Okun MS, Opri E, Cernera S, Molina R, Foote KD, Gunduz A. Differentiating tic electrophysiology from voluntary movement in the human thalamocortical circuit. J Neurol Neurosurg Psychiatry. 2020 May;91(5):533-539. doi: 10.1136/jnnp-2019-321973. Epub 2020 Mar 5. PMID 32139653
- [Background] Bohlhalter S, Goldfine A, Matteson S, Garraux G, Hanakawa T, Kansaku K, Wurzman R, Hallett M. Neural correlates of tic generation in Tourette syndrome: an event-related functional MRI study. Brain. 2006 Aug;129(Pt 8):2029-37. doi: 10.1093/brain/awl050. Epub 2006 Mar 6. PMID 16520330
- [Background] Wang Z, Maia TV, Marsh R, Colibazzi T, Gerber A, Peterson BS. The neural circuits that generate tics in Tourette's syndrome. Am J Psychiatry. 2011 Dec;168(12):1326-37. doi: 10.1176/appi.ajp.2011.09111692. Epub 2011 Sep 28. PMID 21955933
- [Background] Johnson KA, Duffley G, Foltynie T, Hariz M, Zrinzo L, Joyce EM, Akram H, Servello D, Galbiati TF, Bona A, Porta M, Meng FG, Leentjens AFG, Gunduz A, Hu W, Foote KD, Okun MS, Butson CR. Basal Ganglia Pathways Associated With Therapeutic Pallidal Deep Brain Stimulation for Tourette Syndrome. Biol Psychiatry Cogn Neurosci Neuroimaging. 2021 Oct;6(10):961-972. doi: 10.1016/j.bpsc.2020.11.005. Epub 2020 Nov 24. PMID 33536144
- [Background] Johnson KA, Fletcher PT, Servello D, Bona A, Porta M, Ostrem JL, Bardinet E, Welter ML, Lozano AM, Baldermann JC, Kuhn J, Huys D, Foltynie T, Hariz M, Joyce EM, Zrinzo L, Kefalopoulou Z, Zhang JG, Meng FG, Zhang C, Ling Z, Xu X, Yu X, Smeets AY, Ackermans L, Visser-Vandewalle V, Mogilner AY, Pourfar MH, Almeida L, Gunduz A, Hu W, Foote KD, Okun MS, Butson CR. Image-based analysis and long-term clinical outcomes of deep brain stimulation for Tourette syndrome: a multisite study. J Neurol Neurosurg Psychiatry. 2019 Oct;90(10):1078-1090. doi: 10.1136/jnnp-2019-320379. Epub 2019 May 25. PMID 31129620
- [Background] Frey J, Malaty IA. Tourette Syndrome Treatment Updates: a Review and Discussion of the Current and Upcoming Literature. Curr Neurol Neurosci Rep. 2022 Feb;22(2):123-142. doi: 10.1007/s11910-022-01177-8. Epub 2022 Feb 2. PMID 35107785
- [Background] Gao Y, Wang S, Wang A, Fan S, Ge Y, Wang H, Gao D, Wang J, Mao Z, Zhao H, Zhang H, Shi L, Liu H, Zhu G, Yang A, Bai Y, Zhang X, Liu C, Wang Q, Li R, Liang K, Brown KG, Cui Z, Han C, Zhang J, Meng F. Comparison of children and adults in deep brain stimulation for Tourette Syndrome: a large-scale multicenter study of 102 cases with long-term follow-up. BMC Med. 2024 May 30;22(1):218. doi: 10.1186/s12916-024-03432-w. PMID 38816877
- [Background] Schrock LE, Mink JW, Woods DW, Porta M, Servello D, Visser-Vandewalle V, Silburn PA, Foltynie T, Walker HC, Shahed-Jimenez J, Savica R, Klassen BT, Machado AG, Foote KD, Zhang JG, Hu W, Ackermans L, Temel Y, Mari Z, Changizi BK, Lozano A, Auyeung M, Kaido T, Agid Y, Welter ML, Khandhar SM, Mogilner AY, Pourfar MH, Walter BL, Juncos JL, Gross RE, Kuhn J, Leckman JF, Neimat JA, Okun MS; Tourette Syndrome Association International Deep Brain Stimulation (DBS) Database and Registry Study Group. Tourette syndrome deep brain stimulation: a review and updated recommendations. Mov Disord. 2015 Apr;30(4):448-71. doi: 10.1002/mds.26094. Epub 2014 Dec 5. PMID 25476818
- [Background] Baldermann JC, Schuller T, Huys D, Becker I, Timmermann L, Jessen F, Visser-Vandewalle V, Kuhn J. Deep Brain Stimulation for Tourette-Syndrome: A Systematic Review and Meta-Analysis. Brain Stimul. 2016 Mar-Apr;9(2):296-304. doi: 10.1016/j.brs.2015.11.005. Epub 2015 Dec 29. PMID 26827109
- [Background] Jafari F, Abbasi P, Rahmati M, Hodhodi T, Kazeminia M. Systematic Review and Meta-Analysis of Tourette Syndrome Prevalence; 1986 to 2022. Pediatr Neurol. 2022 Dec;137:6-16. doi: 10.1016/j.pediatrneurol.2022.08.010. Epub 2022 Sep 5. PMID 36182698
- [Background] Liu ZS, Cui YH, Sun D, Lu Q, Jiang YW, Jiang L, Wang JQ, Luo R, Fang F, Zhou SZ, Wang Y, Cai FC, Lin Q, Xiong L, Zheng Y, Qin J. Current Status, Diagnosis, and Treatment Recommendation for Tic Disorders in China. Front Psychiatry. 2020 Aug 13;11:774. doi: 10.3389/fpsyt.2020.00774. eCollection 2020. PMID 32903695
- [Background] Hirschtritt ME, Lee PC, Pauls DL, Dion Y, Grados MA, Illmann C, King RA, Sandor P, McMahon WM, Lyon GJ, Cath DC, Kurlan R, Robertson MM, Osiecki L, Scharf JM, Mathews CA; Tourette Syndrome Association International Consortium for Genetics. Lifetime prevalence, age of risk, and genetic relationships of comorbid psychiatric disorders in Tourette syndrome. JAMA Psychiatry. 2015 Apr;72(4):325-33. doi: 10.1001/jamapsychiatry.2014.2650. PMID 25671412
- [Background] Johnson KA, Worbe Y, Foote KD, Butson CR, Gunduz A, Okun MS. Tourette syndrome: clinical features, pathophysiology, and treatment. Lancet Neurol. 2023 Feb;22(2):147-158. doi: 10.1016/S1474-4422(22)00303-9. Epub 2022 Oct 28. PMID 36354027